CLINICAL TRIAL: NCT00399490
Title: OPEN-LABEL, MULTIPLE-DOSE STUDY OF THE SAFETY AND EFFICACY OF RN624 IN ADULTS WITH PAIN DUE TO OSTEOARTHRITIS OF THE KNEE.
Brief Title: Open-label Extension Study Of RN624
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4091009; RN624-CL007 (Other: Alias Study Number)
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis; OA Knee Pain; Arthritis
Keywords: Monoclonal antibody
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — tanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RN624 (PF-04383119)

INTERVENTIONS:
Drug: RN624 (PF-04383119) — 50 mcg/kg

SUMMARY:
Study RN624-CL007 is planned to be an open-label protocol to enroll subjects who have previously participated in Study No. RN624-CL006. In this study, subjects will receive RN624 on an open-label basis.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Study RN624-CL006

Exclusion Criteria:

* The occurrence of any adverse event or condition during the controlled studies that, in the opinion of the Investigator, should exclude the subject from participating in the open-label extension
* Pregnant or lactating female subjects or subjects who do not agree to use an appropriate form of birth control throughout the study and for 3 months after completing the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-09-15 (Actual); Primary Completion 2008-02-11 (Actual); Study Completion 2008-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - BrookWood Internal Medicine, Birmingham, Alabama
  - Radiant Research, Birmingham, Alabama
  - Arizona Research Center, LLC, Phoenix, Arizona
  - Imaging Centers of Anaheim, Anaheim, California
  - Orange County Clinical Research, Anaheim, California
  - Synergy Clinical Research Center, National City, California
  - David M. Radin, MD, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Covance Clinical Research Unit, Inc, Daytona Beach, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - Habana Hospital Pharmacy, Tampa, Florida
  - Covance Clinical Research Unit, Inc. Honolulu, Honolulu, Hawaii
  - Covance Boise, Boise, Idaho
  - Northwest Indiana Center for Clinical Research, Merrillville, Indiana
  - Office of David Neustadt, PSL, Louisville, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Quality Clincal Research, Omaha, Nebraska
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - AAIR Research Center, Rochester, New York
  - Sports Medicine and Orthopaedics Center, Greensboro, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Pharmacotherapy Research Associates Incorporated, Zanesville, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Office of Walter F. Chase, MD, PA, Austin, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Rheumatology Associates of South Texas, San Antonio, Texas
  - South Texas Radiology Imaging Center, San Antonio, Texas
  - Pivotal Research, Midvale, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Clinical Trials Northwest, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schnitzer TJ, Lane NE, Birbara C, Smith MD, Simpson SL, Brown MT. Long-term open-label study of tanezumab for moderate to severe osteoarthritic knee pain. Osteoarthritis Cartilage. 2011 Jun;19(6):639-46. doi: 10.1016/j.joca.2011.01.009. Epub 2011 Jan 18. PMID 21251985
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091009&StudyName=Open-label%20Extension%20Study%20Of%20RN624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had received at least 2 infusions of study drug and had been followed for 56 days after the last infusion in previous study A4091008 (NCT00394563) were eligible to be enrolled in this study.
Groups:
- Tanezumab 50 mcg/kg: Participants who had previously received either tanezumab (RN624 or PF-04383119) 10, 25, 50, 100 or 200 microgram per kilogram (mcg/kg) intravenous infusion or placebo matched to tanezumab infusion in parent study A4091008 (NCT00394563), received tanezumab 50 mcg/kg intravenous infusion over 5 minutes at Day 1 and 56. Additional doses of tanezumab 50 mcg/kg intravenous infusion over 5 minutes at 8 week intervals from Day 56 as per investigator's discretion.
Period: Overall Study
Arm/Group | Tanezumab 50 mcg/kg
Started | 281
Completed | 183
Not Completed | 98
Not completed — Adverse Event | 19
Not completed — Lack of Efficacy | 31
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 18
Not completed — Other | 25

BASELINE CHARACTERISTICS:
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE: an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 12 weeks after last dose that were absent before treatment in this study or that worsened relative to pretreatment state. AEs included both SAEs and non-serious adverse events.
Time Frame: Baseline up to 12 weeks after last dose of study drug
Population: Safety population included all participants who had received at least 1 study drug infusion in this study, A4091009 (NCT00399490).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 281
Participants
  AEs | 168
  SAEs | 8

2. Secondary Outcome: Change From A4091008 (NCT00394563) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from the five individual questions scored on a visual analog scale (VAS) of 0 to 100, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 100, where higher scores indicate higher pain.
Time Frame: A4091008: Baseline, A4091009: Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: Intent-to-treat (ITT) population included all participants who received at least 1 study drug infusion (in this study,A4091009[NCT00399490]) and had at least 1 evaluation post infusion. Here, "overall number of participants analyzed" signifies participants evaluable for this OM and "number analyzed" signifies participants evaluable at each specified row.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tanezumab 50 mcg/kg (Previous Tanezumab Treatment): Participants who had previously received tanezumab 10, 25, 50, 100 or 200 microgram per kilogram (mcg/kg) intravenous infusion in parent study A4091008 (NCT00394563), received tanezumab 50 mcg/kg intravenous infusion over 5 minutes at Day 1 and 56. Additional doses of tanezumab 50 mcg/kg intravenous infusion over 5 minutes at 8 week intervals from Day 56 as per investigator's discretion.
- Tanezumab 50 mcg/kg (Previous Placebo Treatment): Participants who had previously received placebo matched to tanezumab intravenous infusion in parent study A4091008, received tanezumab 50 mcg/kg intravenous infusion over 5 minutes at Day 1 and 56. Additional doses of tanezumab 50 mcg/kg intravenous infusion over 5 minutes at 8 week intervals from Day 56 as per investigator's discretion.
Arm/Group | Tanezumab 50 mcg/kg (Previous Tanezumab Treatment) | Tanezumab 50 mcg/kg (Previous Placebo Treatment)
Number analyzed (Participants) | 236 | 40
units on a scale
  Baseline | 67.4 (12.44) | 67.4 (11.04)
  Change at Week 0: number analyzed (Participants) | 230 | 37
  Change at Week 0 | -25.3 (25.68) | -16.6 (24.21)
  Change at Week 4: number analyzed (Participants) | 221 | 38
  Change at Week 4 | -38.0 (24.54) | -39.1 (21.93)
  Change at Week 8: number analyzed (Participants) | 212 | 39
  Change at Week 8 | -35.9 (24.68) | -34.1 (24.04)
  Change at Week 16: number analyzed (Participants) | 183 | 29
  Change at Week 16 | -33.5 (25.47) | -37.3 (21.42)
  Change at Week 24: number analyzed (Participants) | 148 | 27
  Change at Week 24 | -30.6 (26.31) | -34.0 (22.36)
  Change at Week 32: number analyzed (Participants) | 110 | 22
  Change at Week 32 | -35.4 (24.25) | -27.8 (23.12)
  Change at Week 40: number analyzed (Participants) | 66 | 20
  Change at Week 40 | -27.9 (25.10) | -28.5 (24.91)
  Change at Week 48: number analyzed (Participants) | 42 | 14
  Change at Week 48 | -25.0 (22.86) | -26.3 (23.91)
  Change at Week 56: number analyzed (Participants) | 24 | 8
  Change at Week 56 | -17.2 (23.82) | -22.4 (22.32)
  Change at Week 64: number analyzed (Participants) | 14 | 4
  Change at Week 64 | -18.6 (24.92) | -9.7 (28.70)
  Change at Week 72: number analyzed (Participants) | 2 | 2
  Change at Week 72 | -15.6 (31.40) | -28.3 (5.23)

3. Secondary Outcome: Change From A4091008 (NCT00394563) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in index joint during past 48 hours. It is calculated as mean of the scores from the 2 individual questions scored on VAS of 0 to 100, where higher scores indicate worse function. Total score range for WOMAC stiffness subscale score is 0 to 100, where higher scores indicate worse function. Stiffness is defined as a sensation of decreased ease in movement of knee.
Time Frame: A4091008: Baseline, A4091009: Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: ITT population included all participants who received at least 1 study drug infusion (in this study, A4091009 [NCT00399490]) and had at least 1 evaluation post infusion. Here, "overall number of participants analyzed" signifies participants evaluable for this OM and "number analyzed" signifies participants evaluable at each specified row.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg (Previous Tanezumab Treatment) | Tanezumab 50 mcg/kg (Previous Placebo Treatment)
Number analyzed (Participants) | 236 | 40
units on a scale
  Baseline | 71.9 (15.21) | 71.6 (13.65)
  Change at Week 0: number analyzed (Participants) | 230 | 37
  Change at Week 0 | -25.0 (27.92) | -17.4 (24.27)
  Change at Week 4: number analyzed (Participants) | 221 | 38
  Change at Week 4 | -40.8 (26.19) | -42.2 (21.35)
  Change at Week 8: number analyzed (Participants) | 212 | 39
  Change at Week 8 | -38.9 (27.50) | -36.6 (25.45)
  Change at Week 16: number analyzed (Participants) | 183 | 29
  Change at Week 16 | -34.0 (27.61) | -39.7 (23.93)
  Change at Week 24: number analyzed (Participants) | 148 | 27
  Change at Week 24 | -33.2 (28.97) | -34.7 (24.47)
  Change at Week 32: number analyzed (Participants) | 110 | 22
  Change at Week 32 | -38.1 (26.20) | -26.6 (24.27)
  Change at Week 40: number analyzed (Participants) | 66 | 20
  Change at Week 40 | -27.7 (30.94) | -33.0 (26.57)
  Change at Week 48: number analyzed (Participants) | 42 | 14
  Change at Week 48 | -28.6 (27.59) | -26.6 (24.58)
  Change at Week 56: number analyzed (Participants) | 24 | 8
  Change at Week 56 | -18.7 (25.96) | -22.6 (20.67)
  Change at Week 64: number analyzed (Participants) | 14 | 4
  Change at Week 64 | -22.0 (29.82) | -8.1 (33.04)
  Change at Week 72: number analyzed (Participants) | 2 | 2
  Change at Week 72 | -12.8 (26.52) | -19.0 (14.14)

4. Secondary Outcome: Change From A4091008 (NCT00394563) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint during past 48 hours. It is calculated as the mean of the scores from the 17 individual questions scored on VAS of 0 to 100, where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 to 100, where higher scores indicate worse function.
Time Frame: A4091008: Baseline, A4091009: Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg (Previous Tanezumab Treatment) | Tanezumab 50 mcg/kg (Previous Placebo Treatment)
Number analyzed (Participants) | 236 | 40
units on a scale
  Baseline | 66.7 (13.79) | 67.6 (13.30)
  Change at Week 0: number analyzed (Participants) | 230 | 37
  Change at Week 0 | -24.3 (25.04) | -15.9 (22.04)
  Change at Week 4: number analyzed (Participants) | 221 | 38
  Change at Week 4 | -37.9 (23.94) | -40.2 (20.28)
  Change at Week 8: number analyzed (Participants) | 212 | 39
  Change at Week 8 | -35.4 (24.18) | -34.9 (23.10)
  Change at Week 16: number analyzed (Participants) | 183 | 29
  Change at Week 16 | -32.5 (24.57) | -38.1 (23.72)
  Change at Week 24: number analyzed (Participants) | 148 | 27
  Change at Week 24 | -29.1 (24.62) | -33.0 (23.45)
  Change at Week 32: number analyzed (Participants) | 110 | 22
  Change at Week 32 | -33.3 (24.29) | -27.1 (23.95)
  Change at Week 40: number analyzed (Participants) | 66 | 20
  Change at Week 40 | -26.8 (26.05) | -30.3 (22.71)
  Change at Week 48: number analyzed (Participants) | 42 | 14
  Change at Week 48 | -24.1 (24.55) | -23.6 (23.16)
  Change at Week 56: number analyzed (Participants) | 24 | 8
  Change at Week 56 | -14.1 (24.62) | -22.7 (20.35)
  Change at Week 64: number analyzed (Participants) | 14 | 4
  Change at Week 64 | -20.7 (23.80) | -7.8 (28.39)
  Change at Week 72: number analyzed (Participants) | 2 | 2
  Change at Week 72 | -8.6 (19.42) | -21.4 (4.66)

5. Secondary Outcome: Change From A4091008 (NCT00394563) Baseline Visual Analog Scale (VAS) for Pain Intensity in the Index Knee at Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: Participants answered: "In the past 24 hours, how much pain have you had in your index knee caused by your osteoarthritis?" Participants responded by using a VAS of 0 to 100, where 0 = no pain and 100 = extreme pain, higher scores indicated more pain.
Time Frame: A4091008: Baseline, A4091009: Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg (Previous Tanezumab Treatment) | Tanezumab 50 mcg/kg (Previous Placebo Treatment)
Number analyzed (Participants) | 237 | 40
units on a scale
  Baseline | 69.8 (10.13) | 68.5 (9.65)
  Change at Week 0: number analyzed (Participants) | 230 | 37
  Change at Week 0 | -22.0 (27.46) | -13.0 (26.84)
  Change at Week 4: number analyzed (Participants) | 221 | 38
  Change at Week 4 | -36.5 (25.59) | -39.6 (22.31)
  Change at Week 8: number analyzed (Participants) | 212 | 39
  Change at Week 8 | -34.5 (27.93) | -31.8 (27.06)
  Change at Week 16: number analyzed (Participants) | 183 | 29
  Change at Week 16 | -30.2 (28.43) | -36.9 (24.88)
  Change at Week 24: number analyzed (Participants) | 148 | 27
  Change at Week 24 | -28.5 (29.77) | -29.6 (27.95)
  Change at Week 32: number analyzed (Participants) | 110 | 22
  Change at Week 32 | -32.2 (29.29) | -21.2 (28.05)
  Change at Week 40: number analyzed (Participants) | 66 | 20
  Change at Week 40 | -26.6 (30.78) | -27.1 (25.13)
  Change at Week 48: number analyzed (Participants) | 42 | 14
  Change at Week 48 | -22.5 (27.30) | -25.2 (29.83)
  Change at Week 56: number analyzed (Participants) | 24 | 8
  Change at Week 56 | -14.0 (30.20) | -8.7 (28.32)
  Change at Week 64: number analyzed (Participants) | 14 | 4
  Change at Week 64 | -16.4 (32.61) | -10.8 (36.99)
  Change at Week 72: number analyzed (Participants) | 2 | 2
  Change at Week 72 | -8.4 (17.15) | -29.0 (24.63)

6. Secondary Outcome: Change From A4091008 (NCT00394563) Baseline in Participant Global Assessment Score at Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a VAS of 0 to 100, where 0 = very poor and 100 = very good, where higher scores indicated better health condition.
Time Frame: A4091008: Baseline, A4091009: Week 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg (Previous Tanezumab Treatment) | Tanezumab 50 mcg/kg (Previous Placebo Treatment)
Number analyzed (Participants) | 236 | 40
units on a scale
  Baseline | 53.3 (19.79) | 50.5 (19.63)
  Change at Week 0: number analyzed (Participants) | 230 | 37
  Change at Week 0 | 10.4 (26.33) | 8.4 (20.32)
  Change at Week 4: number analyzed (Participants) | 221 | 38
  Change at Week 4 | 20.3 (29.16) | 25.9 (24.54)
  Change at Week 8: number analyzed (Participants) | 212 | 39
  Change at Week 8 | 18.5 (28.28) | 21.7 (26.28)
  Change at Week 16: number analyzed (Participants) | 183 | 29
  Change at Week 16 | 15.7 (28.66) | 18.2 (31.85)
  Change at Week 24: number analyzed (Participants) | 148 | 27
  Change at Week 24 | 11.1 (30.83) | 10.9 (33.93)
  Change at Week 32: number analyzed (Participants) | 110 | 22
  Change at Week 32 | 15.9 (30.33) | 6.5 (28.76)
  Change at Week 40: number analyzed (Participants) | 66 | 20
  Change at Week 40 | 11.1 (31.18) | 4.2 (29.16)
  Change at Week 48: number analyzed (Participants) | 42 | 14
  Change at Week 48 | 6.7 (25.51) | 7.5 (26.41)
  Change at Week 56: number analyzed (Participants) | 24 | 8
  Change at Week 56 | -8.0 (32.85) | 6.6 (18.94)
  Change at Week 64: number analyzed (Participants) | 14 | 4
  Change at Week 64 | 9.4 (22.87) | 0.8 (30.05)
  Change at Week 72: number analyzed (Participants) | 2 | 2
  Change at Week 72 | 5.0 (12.73) | 25.5 (17.68)

7. Secondary Outcome: Number of Participants With Response to Participant Satisfaction Questionnaire
Description: Participants answered: "Overall, how satisfied are you with the study drug treatment you received as part of this study?" Participants responded by selecting the most appropriate among the following responses: not at all satisfied, a little satisfied, somewhat satisfied, and very satisfied.
Time Frame: A4091009: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 267
Participants
  Baseline: Very Satisfied | 191
  Baseline: Somewhat Satisfied | 36
  Baseline: A Little Satisfied | 14
  Baseline: Not at all Satisfied | 26
  Week 4: Very Satisfied: number analyzed (Participants) | 259
  Week 4: Very Satisfied | 189
  Week 4: Somewhat Satisfied: number analyzed (Participants) | 259
  Week 4: Somewhat Satisfied | 57
  Week 4: A Little Satisfied: number analyzed (Participants) | 259
  Week 4: A Little Satisfied | 11
  Week 4: Not at all Satisfied: number analyzed (Participants) | 259
  Week 4: Not at all Satisfied | 2
  Week 8: Very Satisfied: number analyzed (Participants) | 251
  Week 8: Very Satisfied | 204
  Week 8: Somewhat Satisfied: number analyzed (Participants) | 251
  Week 8: Somewhat Satisfied | 35
  Week 8: A Little Satisfied: number analyzed (Participants) | 251
  Week 8: A Little Satisfied | 9
  Week 8: Not at all Satisfied: number analyzed (Participants) | 251
  Week 8: Not at all Satisfied | 3
  Week 16: Very Satisfied: number analyzed (Participants) | 211
  Week 16: Very Satisfied | 162
  Week 16: Somewhat Satisfied: number analyzed (Participants) | 211
  Week 16: Somewhat Satisfied | 36
  Week 16: A Little Satisfied: number analyzed (Participants) | 211
  Week 16: A Little Satisfied | 12
  Week 16: Not at all Satisfied: number analyzed (Participants) | 211
  Week 16: Not at all Satisfied | 1
  Week 24: Very Satisfied: number analyzed (Participants) | 175
  Week 24: Very Satisfied | 139
  Week 24: Somewhat Satisfied: number analyzed (Participants) | 175
  Week 24: Somewhat Satisfied | 27
  Week 24: A Little Satisfied: number analyzed (Participants) | 175
  Week 24: A Little Satisfied | 8
  Week 24: Not at all Satisfied: number analyzed (Participants) | 175
  Week 24: Not at all Satisfied | 1
  Week 32: Very Satisfied: number analyzed (Participants) | 132
  Week 32: Very Satisfied | 105
  Week 32: Somewhat Satisfied: number analyzed (Participants) | 132
  Week 32: Somewhat Satisfied | 21
  Week 32: A Little Satisfied: number analyzed (Participants) | 132
  Week 32: A Little Satisfied | 5
  Week 32: Not at all Satisfied: number analyzed (Participants) | 132
  Week 32: Not at all Satisfied | 1
  Week 40: Very Satisfied: number analyzed (Participants) | 86
  Week 40: Very Satisfied | 72
  Week 40: Somewhat Satisfied: number analyzed (Participants) | 86
  Week 40: Somewhat Satisfied | 10
  Week 40: A Little Satisfied: number analyzed (Participants) | 86
  Week 40: A Little Satisfied | 3
  Week 40: Not at all Satisfied: number analyzed (Participants) | 86
  Week 40: Not at all Satisfied | 1
  Week 48: Very Satisfied: number analyzed (Participants) | 56
  Week 48: Very Satisfied | 46
  Week 48: Somewhat Satisfied: number analyzed (Participants) | 56
  Week 48: Somewhat Satisfied | 7
  Week 48: A Little Satisfied: number analyzed (Participants) | 56
  Week 48: A Little Satisfied | 3
  Week 48: Not at all Satisfied: number analyzed (Participants) | 56
  Week 48: Not at all Satisfied | 0
  Week 56: Very Satisfied: number analyzed (Participants) | 32
  Week 56: Very Satisfied | 27
  Week 56: Somewhat Satisfied: number analyzed (Participants) | 32
  Week 56: Somewhat Satisfied | 3
  Week 56: A Little Satisfied: number analyzed (Participants) | 32
  Week 56: A Little Satisfied | 2
  Week 56: Not at all Satisfied: number analyzed (Participants) | 32
  Week 56: Not at all Satisfied | 0
  Week 64: Very Satisfied: number analyzed (Participants) | 18
  Week 64: Very Satisfied | 16
  Week 64: Somewhat Satisfied: number analyzed (Participants) | 18
  Week 64: Somewhat Satisfied | 2
  Week 64: A Little Satisfied: number analyzed (Participants) | 18
  Week 64: A Little Satisfied | 0
  Week 64: Not at all Satisfied: number analyzed (Participants) | 18
  Week 64: Not at all Satisfied | 0
  Week 72: Very Satisfied: number analyzed (Participants) | 4
  Week 72: Very Satisfied | 4
  Week 72: Somewhat Satisfied: number analyzed (Participants) | 4
  Week 72: Somewhat Satisfied | 0
  Week 72: A Little Satisfied: number analyzed (Participants) | 4
  Week 72: A Little Satisfied | 0
  Week 72: Not at all Satisfied: number analyzed (Participants) | 4
  Week 72: Not at all Satisfied | 0

8. Secondary Outcome: Change From A4091009 (NCT00399490) Baseline in 36-Item Short-Form Health Survey (SF-36) at Week 4, 8, 16, 24, 32, 40, 48, 56, 64 and 72
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores (CS). The total score for each section and 2 component scores are an average of the individual question scores, which are scaled from 0 to 100, where 0=lowest level of functioning and 100=highest level of functioning, higher scores indicated better functioning .
Time Frame: A4091009: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 271
units on a scale
  Baseline: General Health | 75.9 (16.97)
  Baseline: Physical Function | 45.4 (21.40)
  Baseline: Role Physical | 63.3 (23.61)
  Baseline: Bodily Pain | 50.4 (19.86)
  Baseline: Vitality | 63.2 (18.24)
  Baseline: Social Functioning | 83.9 (19.88)
  Baseline: Role Emotional | 81.3 (22.54)
  Baseline: Mental Health | 82.8 (13.45)
  Change at Week 4: General Health: number analyzed (Participants) | 259
  Change at Week 4: General Health | 3.5 (17.08)
  Change at Week 4: Physical Function: number analyzed (Participants) | 259
  Change at Week 4: Physical Function | 10.4 (19.09)
  Change at Week 4: Role Physical: number analyzed (Participants) | 259
  Change at Week 4: Role Physical | 9.8 (21.45)
  Change at Week 4: Bodily Pain: number analyzed (Participants) | 259
  Change at Week 4: Bodily Pain | 11.3 (22.90)
  Change at Week 4: Vitality: number analyzed (Participants) | 259
  Change at Week 4: Vitality | 6.4 (18.47)
  Change at Week 4: Social Function: number analyzed (Participants) | 259
  Change at Week 4: Social Function | 6.6 (23.29)
  Change at Week 4: Role Emotional: number analyzed (Participants) | 259
  Change at Week 4: Role Emotional | 6.3 (23.09)
  Change at Week 4: Mental Health: number analyzed (Participants) | 259
  Change at Week 4: Mental Health | 4.8 (20.39)
  Change at Week 8: General Health: number analyzed (Participants) | 251
  Change at Week 8: General Health | 3.5 (18.02)
  Change at Week 8: Physical Function: number analyzed (Participants) | 251
  Change at Week 8: Physical Function | 8.6 (19.39)
  Change at Week 8: Role Physical: number analyzed (Participants) | 251
  Change at Week 8: Role Physical | 6.7 (20.15)
  Change at Week 8: Bodily Pain: number analyzed (Participants) | 251
  Change at Week 8: Bodily Pain | 10.9 (22.11)
  Change at Week 8: Vitality: number analyzed (Participants) | 251
  Change at Week 8: Vitality | 4.4 (18.51)
  Change at Week 8: Social Function: number analyzed (Participants) | 251
  Change at Week 8: Social Function | 5.1 (22.41)
  Change at Week 8: Role Emotional: number analyzed (Participants) | 251
  Change at Week 8: Role Emotional | 5.0 (22.87)
  Change at Week 8: Mental Health: number analyzed (Participants) | 251
  Change at Week 8: Mental Health | 4.3 (19.11)
  Change at Week 16: General Health: number analyzed (Participants) | 212
  Change at Week 16: General Health | 2.4 (17.10)
  Change at Week 16: Physical Function: number analyzed (Participants) | 212
  Change at Week 16: Physical Function | 7.8 (20.79)
  Change at Week 16: Role Physical: number analyzed (Participants) | 212
  Change at Week 16: Role Physical | 5.0 (22.86)
  Change at Week 16: Bodily Pain: number analyzed (Participants) | 212
  Change at Week 16: Bodily Pain | 8.5 (24.93)
  Change at Week 16: Vitality: number analyzed (Participants) | 212
  Change at Week 16: Vitality | 3.7 (19.59)
  Change at Week 16: Social Function: number analyzed (Participants) | 212
  Change at Week 16: Social Function | 4.4 (24.04)
  Change at Week 16: Role Emotional: number analyzed (Participants) | 212
  Change at Week 16: Role Emotional | 3.4 (23.24)
  Change at Week 16: Mental Health: number analyzed (Participants) | 212
  Change at Week 16: Mental Health | 1.4 (19.21)
  Change at Week 24: General Health: number analyzed (Participants) | 175
  Change at Week 24: General Health | 2.4 (20.82)
  Change at Week 24: Physical Function: number analyzed (Participants) | 175
  Change at Week 24: Physical Function | 6.6 (21.49)
  Change at Week 24: Role Physical: number analyzed (Participants) | 175
  Change at Week 24: Role Physical | 4.2 (24.74)
  Change at Week 24: Bodily Pain: number analyzed (Participants) | 175
  Change at Week 24: Bodily Pain | 6.1 (26.06)
  Change at Week 24: Vitality: number analyzed (Participants) | 175
  Change at Week 24: Vitality | 4.3 (21.18)
  Change at Week 24: Social Function: number analyzed (Participants) | 175
  Change at Week 24: Social Function | 4.9 (28.94)
  Change at Week 24: Role Emotional: number analyzed (Participants) | 175
  Change at Week 24: Role Emotional | 4.2 (27.76)
  Change at Week 24: Mental Health: number analyzed (Participants) | 175
  Change at Week 24: Mental Health | 3.4 (23.40)
  Change at Week 32: General Health: number analyzed (Participants) | 132
  Change at Week 32: General Health | 1.8 (16.68)
  Change at Week 32: Physical Function: number analyzed (Participants) | 132
  Change at Week 32: Physical Function | 4.3 (22.67)
  Change at Week 32: Role Physical: number analyzed (Participants) | 132
  Change at Week 32: Role Physical | 0.6 (27.42)
  Change at Week 32: Bodily Pain: number analyzed (Participants) | 132
  Change at Week 32: Bodily Pain | 5.9 (25.26)
  Change at Week 32: Vitality: number analyzed (Participants) | 132
  Change at Week 32: Vitality | -0.7 (21.17)
  Change at Week 32: Social Function: number analyzed (Participants) | 132
  Change at Week 32: Social Function | 1.2 (26.23)
  Change at Week 32: Role Emotional: number analyzed (Participants) | 132
  Change at Week 32: Role Emotional | 1.3 (25.79)
  Change at Week 32: Mental Health: number analyzed (Participants) | 132
  Change at Week 32: Mental Health | 0.9 (20.55)
  Change at Week 40: General Health: number analyzed (Participants) | 86
  Change at Week 40: General Health | 1.2 (20.50)
  Change at Week 40: Physical Function: number analyzed (Participants) | 86
  Change at Week 40: Physical Function | 4.4 (25.87)
  Change at Week 40: Role Physical: number analyzed (Participants) | 86
  Change at Week 40: Role Physical | 3.7 (28.57)
  Change at Week 40: Bodily Pain: number analyzed (Participants) | 86
  Change at Week 40: Bodily Pain | 4.1 (29.75)
  Change at Week 40: Vitality: number analyzed (Participants) | 86
  Change at Week 40: Vitality | 1.7 (25.69)
  Change at Week 40: Social Function: number analyzed (Participants) | 86
  Change at Week 40: Social Function | 3.9 (28.41)
  Change at Week 40: Role Emotional: number analyzed (Participants) | 86
  Change at Week 40: Role Emotional | 0.7 (31.17)
  Change at Week 40: Mental Health: number analyzed (Participants) | 86
  Change at Week 40: Mental Health | 2.2 (24.06)
  Change at Week 48: General Health: number analyzed (Participants) | 56
  Change at Week 48: General Health | 2.2 (22.13)
  Change at Week 48: Physical Function: number analyzed (Participants) | 56
  Change at Week 48: Physical Function | -0.9 (25.28)
  Change at Week 48: Role Physical: number analyzed (Participants) | 56
  Change at Week 48: Role Physical | -5.2 (31.66)
  Change at Week 48: Bodily Pain: number analyzed (Participants) | 56
  Change at Week 48: Bodily Pain | 0.4 (27.77)
  Change at Week 48: Vitality: number analyzed (Participants) | 56
  Change at Week 48: Vitality | -2.8 (24.14)
  Change at Week 48: Social Function: number analyzed (Participants) | 56
  Change at Week 48: Social Function | -2.1 (30.99)
  Change at Week 48: Role Emotional: number analyzed (Participants) | 56
  Change at Week 48: Role Emotional | -5.1 (32.43)
  Change at Week 48: Mental Health: number analyzed (Participants) | 56
  Change at Week 48: Mental Health | 1.4 (24.70)
  Change at Week 56: General Health: number analyzed (Participants) | 32
  Change at Week 56: General Health | -0.5 (19.18)
  Change at Week 56: Physical Function: number analyzed (Participants) | 32
  Change at Week 56: Physical Function | -3.5 (24.90)
  Change at Week 56: Role Physical: number analyzed (Participants) | 32
  Change at Week 56: Role Physical | -6.2 (28.08)
  Change at Week 56: Bodily Pain: number analyzed (Participants) | 32
  Change at Week 56: Bodily Pain | -0.4 (22.64)
  Change at Week 56: Vitality: number analyzed (Participants) | 32
  Change at Week 56: Vitality | -3.9 (21.99)
  Change at Week 56: Social Function: number analyzed (Participants) | 32
  Change at Week 56: Social Function | -4.6 (26.65)
  Change at Week 56: Role Emotional: number analyzed (Participants) | 32
  Change at Week 56: Role Emotional | -6.2 (29.92)
  Change at Week 56: Mental Health: number analyzed (Participants) | 32
  Change at Week 56: Mental Health | -6.2 (21.69)
  Change at Week 64: General Health: number analyzed (Participants) | 18
  Change at Week 64: General Health | 0.5 (23.42)
  Change at Week 64: Physical Function: number analyzed (Participants) | 18
  Change at Week 64: Physical Function | -2.6 (14.27)
  Change at Week 64: Role Physical: number analyzed (Participants) | 18
  Change at Week 64: Role Physical | -1.6 (25.04)
  Change at Week 64: Bodily Pain: number analyzed (Participants) | 18
  Change at Week 64: Bodily Pain | -2.9 (22.13)
  Change at Week 64: Vitality: number analyzed (Participants) | 18
  Change at Week 64: Vitality | -4.4 (24.09)
  Change at Week 64: Social Function: number analyzed (Participants) | 18
  Change at Week 64: Social Function | -0.5 (32.43)
  Change at Week 64: Role Emotional: number analyzed (Participants) | 18
  Change at Week 64: Role Emotional | -2.6 (30.12)
  Change at Week 64: Mental Health: number analyzed (Participants) | 18
  Change at Week 64: Mental Health | 2.1 (26.50)
  Change at Week 72: General Health: number analyzed (Participants) | 4
  Change at Week 72: General Health | -5.0 (4.08)
  Change at Week 72: Physical Function: number analyzed (Participants) | 4
  Change at Week 72: Physical Function | 5.0 (14.72)
  Change at Week 72: Role Physical: number analyzed (Participants) | 4
  Change at Week 72: Role Physical | 0.0 (5.10)
  Change at Week 72: Bodily Pain: number analyzed (Participants) | 4
  Change at Week 72: Bodily Pain | -0.0 (14.63)
  Change at Week 72: Vitality: number analyzed (Participants) | 4
  Change at Week 72: Vitality | -9.4 (10.83)
  Change at Week 72: Social Function: number analyzed (Participants) | 4
  Change at Week 72: Social Function | 6.3 (7.22)
  Change at Week 72: Role Emotional: number analyzed (Participants) | 4
  Change at Week 72: Role Emotional | -10.4 (12.50)
  Change at Week 72: Mental Health: number analyzed (Participants) | 4
  Change at Week 72: Mental Health | -1.3 (9.46)

9. Secondary Outcome: Percentage of Participants Who Discontinued the Study
Time Frame: A4091009: Baseline up to 12 weeks after last dose of study drug
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 281
percentage of participants | 34.9

10. Secondary Outcome: Median Time in Study A4091009
Description: Median time of participation in the study for all the participants was evaluated.
Time Frame: A4091009: Baseline up to 12 weeks after last dose of study drug
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 281
days | 198 [1.0 to 484.0]

11. Other Pre Specified Outcome: Change From A4091009 (NCT00399490) Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score at Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, and End of Study
Description: HVLT-R: instrument consisting of 12 noun list, used to measure verbal learning and memory (recognition and recall). List was read to participant, who then attempted to recall as many words as possible. The examiner recorded each response. Task was repeated 2 more times, for total of 3 learning trials. After delay interval of 20-25 minutes, delayed recall trial was administered. Total score (TS) = sum of 3 learning trial scores of 12 word each, ranged: 0 (no memory) to 36 (best memory), where higher scores indicated better memory. Delayed recall (DR) = number of words recalled in delayed recall test, ranged: 0 (no memory) to 12 (best memory), where higher scores indicated better memory.
Time Frame: A4091009: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, End of Study (12 weeks after the last dose of study drug)
Population: Safety population included all participants who had received at least 1 study drug infusion in this study, A4091009 (NCT00399490). Here, "overall number of participants analyzed" signifies participants evaluable for this OM and "number analyzed" signifies participants evaluable at each specified row.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 50 mcg/kg
Number analyzed (Participants) | 277
units on a scale
  Baseline: TS: number analyzed (Participants) | 276
  Baseline: TS | 31.5 (3.75)
  Baseline: DR: number analyzed (Participants) | 276
  Baseline: DR | 11.2 (1.44)
  Change at Week 4: TS: number analyzed (Participants) | 269
  Change at Week 4: TS | -0.0 (3.44)
  Change at Week 4: DR: number analyzed (Participants) | 269
  Change at Week 4: DR | -0.0 (1.16)
  Change at Week 8: TS: number analyzed (Participants) | 259
  Change at Week 8: TS | -0.2 (3.43)
  Change at Week 8: DR: number analyzed (Participants) | 259
  Change at Week 8: DR | 0.1 (1.45)
  Change at Week 16: TS: number analyzed (Participants) | 214
  Change at Week 16: TS | 0.1 (3.20)
  Change at Week 16: DR: number analyzed (Participants) | 214
  Change at Week 16: DR | 0.1 (1.33)
  Change at Week 24: TS: number analyzed (Participants) | 178
  Change at Week 24: TS | -0.0 (3.78)
  Change at Week 24: DR: number analyzed (Participants) | 178
  Change at Week 24: DR | 0.1 (1.25)
  Change at Week 32: TS: number analyzed (Participants) | 131
  Change at Week 32: TS | 0.6 (3.53)
  Change at Week 32: DR: number analyzed (Participants) | 131
  Change at Week 32: DR | 0.3 (1.29)
  Change at Week 40: TS: number analyzed (Participants) | 86
  Change at Week 40: TS | 1.1 (3.56)
  Change at Week 40: DR: number analyzed (Participants) | 86
  Change at Week 40: DR | 0.4 (1.27)
  Change at Week 48: TS: number analyzed (Participants) | 57
  Change at Week 48: TS | 0.2 (3.82)
  Change at Week 48: DR: number analyzed (Participants) | 57
  Change at Week 48: DR | 0.2 (1.59)
  Change at Week 56: TS: number analyzed (Participants) | 32
  Change at Week 56: TS | -0.0 (3.83)
  Change at Week 56: DR: number analyzed (Participants) | 32
  Change at Week 56: DR | 0.2 (1.47)
  Change at Week 64: TS: number analyzed (Participants) | 19
  Change at Week 64: TS | 1.1 (3.81)
  Change at Week 64: DR: number analyzed (Participants) | 19
  Change at Week 64: DR | 1.4 (2.09)
  Change at Week 72: TS: number analyzed (Participants) | 5
  Change at Week 72: TS | 1.2 (4.15)
  Change at Week 72: DR: number analyzed (Participants) | 5
  Change at Week 72: DR | 0.2 (0.45)
  Change at End of Study: TS | 0.3 (3.48)
  Change at End of Study: DR | 0.2 (1.25)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tanezumab 50 mcg/kg
Serious Adverse Events (participants affected / at risk) | 8/281
Other Adverse Events (participants affected / at risk) | 112/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 50 mcg/kg (N=281)
Myocardial infarction (Cardiac disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Migraine (Nervous system disorders) | 1
Spinal cord ischaemia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 50 mcg/kg (N=281)
Oedema peripheral (General disorders) | 10
Nasopharyngitis (Infections and infestations) | 12
Sinusitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 13
Urinary tract infection (Infections and infestations) | 11
Contusion (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 17
Joint effusion (Musculoskeletal and connective tissue disorders) | 13
Joint swelling (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Synovial cyst (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 16
Hypoaesthesia (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 7

LIMITATIONS AND CAVEATS:
Data for rescue medication was recorded on the concomitant medication page of the case report form (CRF) as 'pro re nata (as needed)' rather than 'as pill counts'; hence total daily dose of rescue medication received was not recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.